CLINICAL TRIAL: NCT06586645
Title: Evaluation of a Brief, Scalable Module to Mitigate Suicidal Ideation Among Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-24-0374
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety Planning and "Give to Others" Module (Experimental): A standard suicide risk assessment and management protocol followed by the "Give to Others" Module which is a brief cognitive behavioral intervention.
  Interventions: Behavioral: Safety Planning; Behavioral: Give to Others Module
- Safety Planning (Active Comparator): A standard suicide risk assessment and management protocol.
  Interventions: Behavioral: Safety Planning

INTERVENTIONS:
Behavioral: Safety Planning — Safety planning is a standard suicide risk assessment and management protocol. This protocol involves determining level of risk based on current and prior suicidal thoughts and behavior, and then collaborative planning with youth and families for self-monitoring, self-regulation, help seeking, and suicide means restriction.
Behavioral: Give to Others Module — The "Give to Others" Module is a brief cognitive behavioral intervention targeting youth burden-related beliefs. It consists of one primary session and brief phone follow-up.
  Arms: Safety Planning and "Give to Others" Module

SUMMARY:
This project is designed to test a brief therapy to reduce suicidal ideation among a diverse sample of youths ages 12 to 17 who experience anxiety or depression. The goal of the study is to conduct a clinical trial testing whether this therapy reduces suicidal ideation and related beliefs that one is a burden on others. This project will contribute to the field by potentially showing evidence supportive of a brief strategy to reduce suicidal ideation in a way that can be readily understood and used by mental health providers in the community.

DETAILED DESCRIPTION:
This project tests the ability of a brief therapy module to engage youth perceived burdensomeness (PB) in a rigorous randomized controlled trial (RCT) of the intervention, the "Give to Others (GO)" module. The investigators will target PB among 60 ethnically/racially diverse clinic-referred youths (ages 12-17) who experience subacute suicide ideation SI (i.e., positive suicide risk screen; stable safety status). Youths will be recruited from the clinical and community settings and will be randomized to one of the following 2 arms: an assessment and suicide risk management condition (Safety Planning control arm); and a Safety Planning plus GO module condition. The investigators hypothesize that youths receiving the GO module will have lower levels of PB at post-treatment compared with youths who receive the control arm. The investigators also hypothesize that youths receiving the GO module will have lower levels of PB at post-treatment compared to pre-treatment levels.

ELIGIBILITY:
Inclusion Criteria

Adolescents must:

* be between ages 12 and 17 years
* score at or above 4 on the Interpersonal Needs Questionnaire- Burdensomeness Scale
* have a positive screen for suicide risk (i.e., endorsement of suicidal ideation via self-report or parent-report).

Exclusion Criteria

For adolescents to be excluded, they must:

* have cognitive impairment or developmental delay which does not allow for the completion of basic study procedures (i.e., reading and filling out questionnaires; talking to a clinician)
* show imminent risk or a history of hurting themselves or others requiring intensive and restrictive services
* be involved currently in a psychosocial treatment

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Interpersonal Needs Questionnaire- Burdensomenes Scale- Self-report | post-intervention (within one week of completing the assigned intervention)
  5-item youth self-ratings on perceived burdensomeness over the past week. Each item is scored 1-7 (1 = not at all true for me; 7 = very true for me), yielding a total between 5 and 35. Higher scores indicate higher levels of perceived burdensomeness (worse outcome).

SECONDARY OUTCOMES:
Interpersonal Needs Questionnaire- Burdensomenes Scale- Parent report | post-intervention (within one week of completing the assigned intervention)
  5-item parent ratings on youth perceived burdensomeness over the past week. Each item is scored 1-7 (1 = not at all true for me; 7 = very true for me), yielding a total between 5 and 35. Higher scores indicate higher levels of perceived burdensomeness (worse outcome).
Sentence Completion Task- Liability Index | post-intervention (within one week of completing the assigned intervention)
  28-item youth completed task assessing burden-related interpretation bias. Participants read 28 sentences indicative of posing a liability on others and select negatively- or positively-valenced words to complete each sentence. Each item is scored 0 or 1, yielding a total score between 0 and 28. Higher scores indicate higher levels of burden interpretation bias (worse outcome).
Sentence Completion Task- Social Contribution Index | post-intervention (within one week of completing the assigned intervention)
  14-item youth completed task assessing contribution-related interpretation bias. Participants read 14 sentences indicative of contributing to others and select negatively- or positively-valenced words to complete each sentence. Each item is scored 0 or 1, yielding a total score between 0 and 14. Higher scores indicate higher levels of contribution interpretation bias (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Victor Buitron, PhD, Principal Investigator — Florida International University
Locations (1):
- FIU Center for Children and Families, Miami, Florida, United States